CLINICAL TRIAL: NCT03524768
Title: Microvascular Endothelial Function in a Cohort of Patients With the Cardiac Form of Chronic Chagas Disease.
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, MD, PhD, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: CHAGASKASALTIBIRIÇÁ
Record Dates: First submitted 2018-04-21; First posted 2018-05-15 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Chagas Cardiomyopathy
Keywords: endothelial function, microvascular; laser speckle contrast imaging; capillaroscopy, skin
MeSH Terms: conditions — Chagas Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients presenting with Chagas cardiomyopathy: Evaluation of systemic microvascular reactivity using laser speckle contrast imaging Evaluation of skin capillary density using video-capillaroscopy
  Interventions: Diagnostic Test: skin laser speckle contrast imaging and video-capillaroscopy
- control group: Evaluation of systemic microvascular reactivity using laser speckle contrast imaging Evaluation of skin capillary density using video-capillaroscopy
  Interventions: Diagnostic Test: skin laser speckle contrast imaging and video-capillaroscopy

INTERVENTIONS:
Diagnostic Test: skin laser speckle contrast imaging and video-capillaroscopy — Evaluation of endothelial-dependent microvascular reactivity and capillary recruitment

SUMMARY:
The present study aims to evaluate the microvascular endothelial function of a single centre cohort of patients with the cardiac form of Chagas disease, and to search for associations with clinical and laboratory variables.

DETAILED DESCRIPTION:
Chagas disease is an endemic anthropozoonosis in South America, caused by the protozoaTrypamosoma cruzi. Between 15 and 17 million people are estimated to be infected by the parasite in South America. During the chronic phase, 30 to 40% of patients develop the cardiac or intestinal forms of the disease. The myocardial involvement is divided in two subtypes, according to the presence or absence of systolic ventricular dysfunction. The first type is characterized by heart failure symptoms. The second is acknowledged by the development of various degrees of atrioventricular blockade and by tachyarrhythmias.

Microcirculation function is recognized as a fundamental aspect in the pathophysiology of cardiovascular diseases. The identification of endothelial dysfunction by techniques that assess the microvasculature is considered as both a progression and prognostic marker in various conditions, including hypertension, coronary heart disease, and heart failure.

The effects of T. cruzi infection in vascular function were evaluated in previous studies, performed in animals with acute infection. Previous studies in humans observed medium size vessels (brachial artery), in small groups of patients, most without cardiac dysfunction. There are no studies evaluating the microcirculation of patients with the cardiac form of Chagas disease.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with Chagas cardiomyopathy

Exclusion Criteria:

* diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The present study aims to evaluate the microvascular endothelial function of a single centre cohort of patients presenting with the cardiac form of Chagas disease in the National Institute of Cardiology, Ministry of Health, Rio de Janeiro,, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependent skin microvascular function | 2 hours
  systemic microvascular vasodilation induced by endothelium-dependent agents

SECONDARY OUTCOMES:
Endothelium-dependent skin capillary density | 1 hour
  capillary opening induced by post-occlusive reactive hyperemia

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided